CLINICAL TRIAL: NCT02755714
Title: Ipratropium Bromide (Atrovent®) Used to Treat Exercise Induced Laryngeal Obstruction (EILO). An Open Label Pilot Study
Brief Title: Atrovent in Exercise Induced Laryngeal Obstruction (EILO)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014/1885
Record Dates: First submitted 2016-04-18; First posted 2016-04-29 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Exercise Induced Laryngeal Obstruction (EILO)
MeSH Terms: interventions — Ipratropium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Atrovent ® (No Intervention): NO INTERVENTION: The patient will not receive Ipratropium bromide spray (MDI) 20 μg ,(Atrovent ®) prior to CLE testing
- Atrovent ® (Experimental): INTERVENTION: Ipratropium bromide spray (MDI) 20 μg (Atrovent ®) prior to CLE testing
  Interventions: Drug: Ipratropium bromide spray

INTERVENTIONS:
Drug: Ipratropium bromide spray — The patient will - or will not - receive Ipratropium bromide spray (MDI) 20 μg given through a plastic spacer two puffs 1 hour before a continuous laryngoscopy exercise test (CLE-test)
  Other Names: Atrovent
  Arms: Atrovent ®

SUMMARY:
Exercise Induced Laryngeal Obstruction (EILO) is a condition not uncommon in otherwise healthy young people. EILO is caused by posteromedial collapse of supraglottic structures or medialization of the vocal folds, or both, during high intensity exercise. There are currently no treatments available that is properly evidence based. However, case reports suggest a possible effect from the "asthma drug" Ipratropium Bromide (Atrovent®). The current project is an open label pilot study, aiming to test if Atrovent can influence the occurence of EILO, either postponing the onset during exercise or fully prevent the condition to occur.

DETAILED DESCRIPTION:
Exercise induced inspiratory symptoms (EIIS) is increasingly recognized as an important differential diagnosis to exercise induced asthma (EIA) in otherwise healthy adolescents. EIIS is most often linked to laryngeal abnormalities and if so, often labelled exercise induced laryngeal obstruction (E-ILO). In unselected populations, E-ILO has been found in 7.5% and 5.7% of adolescents. Causal mechanisms remain unclear, and a variety of structural and/or functional pathways have been proposed, such as abnormalities related to the epiglottis, the laryngeal cartilage-skeleton or its support, mucosal structures as well as the laryngeal muscular system or its nerve supply. All these abnormalities might conceivably disturb the airflow on its way through the laryngeal inlet, increase the turbulence and the airflow resistance, and thereby set up a sense of dyspnea and trigger the symptoms that are characteristic of EIIS. Additionally, various psychological characteristics have been proposed to be implicated in this causal cascade.

As the causal mechanisms of E-ILO have not been clarified, all attempts on treatment of this condition have been empirical and there is currently no properly evidence-based treatment available. Speech therapy, often in combination with some kind of psychotherapy, have been viewed as mainstay therapy by most authors, whereas other psychological measures such as relaxation therapy, hypnosis and biofeedback have been advocated by others. Anticholinergic aerosols applied before exercise has been suggested and there are reports of successful surgical treatment using laser supraglottoplasty. The common goal of these treatment initiatives has been to increase the size of the laryngeal inlet during the increasing airflow velocity that is induced by increasing exercise intensity.

Inducible laryngeal obstructions were previously often labeled vocal cord dysfunction (VCD), and Ayres et al. proposed in 2002 in an article in Thorax that VCD could be a function of an altered autonomic balance. This view opened for a theoretical framework for treatment of VCD using inhaled anticholinergic agents such as Ipratropium bromide (Atrovent®).

To our knowledge, positive effects from inhaled anticholinergic agents in VCD have so far only been published as case reports, and systematic studies have not been performed.

This study aims to address potential effects from Atrovent in patients with E-ILO verified during a continuous laryngoscopy exercise (CLE) test. The study will primarily include 20 patients consecutively referred to our clinic for EIIS and diagnosed with E-ILO during a routine CLE test. Requirement for inclusion will be a CLE score ≥ 3. The primary endpoint will be the laryngeal response to maximal exercise, described quantitatively by a blinded observer using the CLE score system. Two CLE tests will be performed in each subject, one with - and one without - prior treatment with Atrovent. The patient will thus serve as her/his own control. Half the patients will receive Atrovent before the first study test (at T1), the other half before the second (at T2).

The CLE-test

The CLE-test was described in detail by the authors Heimdal et al. in the "Laryngoscope" in 2006 and the scoring system by Maat et al. in the "European Archives of Otorhinolaryngology" in 2009. In short, the test combines a full cardio-pulmonary treadmill exercise set-up with continuous real-time transnasal video-laryngoscopy applied from rest to peak exercise to rest. A camera and a microphone placed in front of the subject enable recording of simultaneous video images of the external upper part of the body as well as recordings of the respiratory sounds. The subjects run on a treadmill according to a standardized protocol, incrementing speed and/or grade every minute with the aim to obtain peak oxygen consumption (peakVO2) after 6-12 min of exercise. The test is considered successful if the patient experience respiratory complaints, or indicate exhaustion, preferably supported by a plateau in oxygen consumption and/or the heart rate. All recordings continue until normal breathing is regained.

The CLE-test scoring system was established based on evaluations of video recordings from both patients and symptom-negative controls who were examined with the CLE-test. The CLE-test scoring system encompasses separate assessments of the extent of medial rotation of the aryepiglottic folds and adduction of the vocal folds scored in representative respiratory cycles at two different points in time during the exercise session; i.e. at a moderate effort (when changing from walking to running on the treadmill) and at maximal effort (shortly before exhaustion). Adduction is graded from 0 (neutral position or abduction) to a maximum score of 3. This set-up establishes four sub-scores ranging from 0 to 3, i.e. glottic and supraglottic adduction at moderate (A and B), and maximal exercise (C and D). The sum score (E) may finally be categorized into three clusters: 0-2 (normal) and 3-4 (moderate) and 5 or more (severe).

The study has been approved by the Western Norway Regional Committee for Medical and Health Research Ethics (REKVEST 2014/1885) and by the Norwegian Medicines Agency; European Union Drug Regulating Authorities Clinical Trials (EUDRACT) No. 2014-000302-34 (enclosed). The study will be performed under the guidance of the Paediatric Clinical Trial Unit at Haukeland University Hospital, a unit that has extensive experience in running clinical trials in children.

ELIGIBILITY:
Inclusion Criteria: Exercise Induced Inspiratory Symptoms and a CLE score Equal to or larger than three Exclusion Criteria: Participants should be free from co-morbidities other than stable and weel treated asthma. Pregnancy

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
CLE test-scores (please se above; Detailed Study Description) | At exhaustion when the test stops, approximately 10-15 minutes after test commencement
  CLE test-scores will be rated from videos obtained during the CLE test

SECONDARY OUTCOMES:
Patient perceived breathing difficulties during the CLE test | At exhaustion when the test stops, approximately 10-15 minutes after test commencement
  At exhaustion when the test stops, approximately 10-15 minutes after commencement
Investigator scored breathing difficulties during the CLE test | At exhaustion when the test stops, approximately 10-15 minutes after test commencement

CONTACTS AND LOCATIONS:
Overall Officials: BERG ANSGAR, MD and PhD, Study Director — HAUKELAND UNIVERSITY HOSPITAL, PEDIATRIC DEPARTMENT
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Roksund OD, Heimdal JH, Olofsson J, Maat RC, Halvorsen T. Larynx during exercise: the unexplored bottleneck of the airways. Eur Arch Otorhinolaryngol. 2015 Sep;272(9):2101-9. doi: 10.1007/s00405-014-3159-3. Epub 2014 Jul 18. PMID 25033930
- [Background] Christopher KL, Wood RP 2nd, Eckert RC, Blager FB, Raney RA, Souhrada JF. Vocal-cord dysfunction presenting as asthma. N Engl J Med. 1983 Jun 30;308(26):1566-70. doi: 10.1056/NEJM198306303082605. PMID 6406891
- [Background] Maat RC, Hilland M, Roksund OD, Halvorsen T, Olofsson J, Aarstad HJ, Heimdal JH. Exercise-induced laryngeal obstruction: natural history and effect of surgical treatment. Eur Arch Otorhinolaryngol. 2011 Oct;268(10):1485-92. doi: 10.1007/s00405-011-1656-1. Epub 2011 Jun 5. PMID 21643933
- [Background] Johansson H, Norlander K, Berglund L, Janson C, Malinovschi A, Nordvall L, Nordang L, Emtner M. Prevalence of exercise-induced bronchoconstriction and exercise-induced laryngeal obstruction in a general adolescent population. Thorax. 2015 Jan;70(1):57-63. doi: 10.1136/thoraxjnl-2014-205738. Epub 2014 Nov 7. PMID 25380758
- [Background] Hull JH, Selby J, Sandhu G. "You say potato, I say potato": time for consensus in exercise-induced laryngeal obstruction? Otolaryngol Head Neck Surg. 2014 Nov;151(5):891-2. doi: 10.1177/0194599814549529. No abstract available. PMID 25344097
- [Result] Muralitharan P, Carlsen P, Hilland M, Delestre-Levai I, Vollsaeter M, Hufthammer KO, Engan M, Roksund OD, Halvorsen T, Clemm HH. Use of inhaled ipratropium bromide to improve exercise-induced laryngeal obstruction cannot be recommended. ERJ Open Res. 2023 Jan 23;9(1):00308-2022. doi: 10.1183/23120541.00308-2022. eCollection 2023 Jan. PMID 36699648